CLINICAL TRIAL: NCT01868321
Title: Practice of Ventilation in Critically Ill Patients Without Acute Respiratory Distress Syndrome - An International Observational Study
Brief Title: Practice of Ventilation in Critically Ill Patients Without ARDS
Acronym: PRoVENT
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Marcus J. Schultz (Other)
Collaborators: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: PRoVENT
Record Dates: First submitted 2013-05-28; First posted 2013-06-04 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Mechanical Ventilation
Keywords: Mechanical ventilation; Acute respiratory failure; Acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mechanical Ventilation: Patients under mechanical ventilation in the ICU

SUMMARY:
The purpose of this international, multicenter study is to determine ventilation practice and outcomes of intubated and ventilated intensive care unit (ICU) patients. Ventilation characteristics and outcomes will be compared between patients without the acute respiratory distress syndrome (ARDS), patients at risk for ARDS, and patients with mild, moderate or severe ARDS.

Participating centres worldwide will include adult patients undergoing mechanical ventilation in the ICU during a 7-day period. Patients data will be collected during the first 7 days in the ICU, or until ICU discharge. Follow up is until day 90. Primary endpoint is the tidal volume size used during mechanical ventilation. Secondary endpoints are development of ARDS in patients without ARDS at the onset of mechanical ventilation, worsening of ARDS in patients with ARDS at the onset of mechanical ventilation, pulmonary infection, other pulmonary complications, need for tracheostomy, extra-pulmonary complications, duration of ventilation, length of ICU and hospital stay, and ICU, hospital and 90-day mortality.

DETAILED DESCRIPTION:
Research questions:

1. Does ventilation practice, in particular tidal volume size, varies amongst patients without ARDS, patients at risk for ARDS, and patients with mild ARDS?
2. Are tidal volumes used in patients without ARDS higher than those used in patients with ARDS?
3. Are the outcomes in patients without ARDS dependent on the size of tidal volumes?

   * Methods: In this international observational study, consecutive patients in the ICU under mechanical ventilation are eligible for participation. Patients in participating centers will be screened on a daily basis. Patients in mechanical ventilation will be included during a 7-day period, from Monday at 8:00 AM to the next Monday at 7:59 AM (in time zones of the participating centers). The inclusion period will be flexible for participating centers and determined at a later stage together with the study-coordinator.

Times points of data collection:

1. Demographic data and baseline data, including severity scores (e.g. APACHE II-scores and SAPS III) and LIPS, are collected from the clinical files on the day of intubation
2. Ventilation settings, gas exchange variables and vital parameters are collected once a daily in the morning, until ventilation is stopped
3. Chest radiography data from available chest X-rays (i.e., no extra chest X-rays are obtained)
4. Predefined complications are recorded from medical chart until discharge from ICU or death, whatever comes first
5. Length of ICU and hospital stay, and ICU, hospital and 90-day mortality

   * Centres: The investigators aim to recruit 40 - 150 centers worldwide.
   * Ethics Approval: National coordinators will be responsible for clarifying the need for ethics approval and applying for this where appropriate according to local policy. Centres will not be permitted to record data unless ethics approval or an equivalent waiver is in place. The investigators expect that in most, if not every participating country, a patient informed consent is not be required.
   * Monitoring: Due to the observational nature of the study, a DSMB is not be necessary.
   * Study Population: Adult patients in the ICU under mechanical ventilation.
   * Data Collection: Data will be collected at inclusion, every day during seven days, day of ICU and hospital discharge and on day 90. Data will be coded by a patient identification number (PIN) of which the code will be kept safe at the local sites. The data will be transcribed by local investigators onto an internet based electronic CRF.
   * Sample Size Calculation: We did not perform a formal sample size calculation, seen the largely descriptive character of this investigation. We expect to collect data from at least 1000 patients, which will be sufficient to test the hypotheses.
   * Statistical Analysis: Patient characteristics will be compared and described by appropriate statistics. Student's t-test or Mann-Whitney U-tests are used to compare continuous variables and chi-squared tests are used for categorical variables. Data are expressed as means (SD), medians (interquartile range) and proportions as appropriate. Comparisons between and within groups are performed using one-way ANOVA and post-hoc analyses for continuous variables.

The primary analysis concerns the determination of (variation of) tidal volume size in patients without ARDS. Tidal volume size is compared between predefined patient groups: patients at no risk for ARDS, patients at risk for ARDS, patients with mild ARDS, and patients with moderate or severe ARDS.

To identify potential factors associated with outcome like development of ARDS, or worsening of ARDS, development of pulmonary complications, duration of ventilation, or death, univariate analyses are performed. A multivariate logistic regression model is used to identify independent risk factors. A stepwise approach is used to enter new terms into the model, with a limit of p < 0.2 to enter the terms. Time to event variables are analyzed using Cox regression and visualized by Kaplan-Meier.

- Organization: The study is conducted by the PROtective VEntilation Network (PROVENet). National co-ordinators will lead the project within individual nations and identify participating hospitals, translate study paperwork, distribute study paperwork and ensure necessary regulatory approvals are in place. They provide assistance to the participating clinical sites in trial management, record keeping and data management. Local coordinators in each site will supervise data collection and ensure adherence to Good Clinical Practice during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a participating ICU
* Intubated in the participating ICU, or in the emergency room or operation room before the present ICU admission

Exclusion Criteria:

* Age < 18 years
* Receiving only non-invasive ventilation
* Patients under invasive mechanical ventilation previous to the 7-day period of inclusion
* Patients transferred from another hospital under invasive mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated and ventilated ICU-patients.
Sampling Method: Probability Sample
Enrollment: 1030 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Tidal Volume Size | During mechanical ventilation
  Tidal volume size in milliliters per kilogram of predicted body weight

SECONDARY OUTCOMES:
Other Ventilation Parameters | During mechanical ventilation
  Plateau and peak pressure, positive end-expiratory pressure, driving pressure, respiratory rate, inspired oxygen fraction, inspiration to expiration ratio, and minute volume
Development of ARDS | From date of inclusion until the date of first documented ARDS or date of hospital discharge or death from any cause, whichever came first, assessed up to three months
  Patients are defined as having ARDS if they met the Berlin criteria for ARDS.
Worsening of ARDS | From date of inclusion until the date of first documented worsening of ARDS or date of hospital discharge or death from any cause, whichever came first, assessed up to three months
  Defined as any worse in the degree of severity according to Berlin criteria.
Other Pulmonary Complications | From date of inclusion until the date of first documented pulmonary complication or date of hospital discharge or death from any cause, whichever came first, assessed up to three months
  Atelectasis, barotrauma, pleural effusion
Pulmonary Infection | From date of inclusion until the date of first documented pulmonary infection or date of hospital discharge or death from any cause, whichever came first, assessed up to three months
  Defined as need of new antibiotics plus at least one of the following criteria: 1) new or changed sputum; 2) new or changed lung opacities on chest X-ray; 3) temperature > 38.3 ºC; or 4) WBC count > 12,000.
Need for Tracheostomy | From date of inclusion until the date of first documented tracheostomy or date of hospital discharge or death from any cause, whichever came first, assessed up to three months
  Need for tracheostomy during hospital stay
Extra-Pulmonary Complications | From date of inclusion until the date of first documented extra-pulmonary complication or date of hospital discharge or death from any cause, whichever came first, assessed up to three months
  Acute kidney injury, circulatory failure, gastrointestinal failure, acute or exacerbation of chronic heart failure, liver failure, and delirium.
Duration of Mechanical Ventilation | During mechanical ventilation
  Time between orotracheal intubation and successful extubation; note: in case of intermittent MV via a tracheostomy, every day a patient needs MV counts as one extra day of MV, irrespective of duration of MV that specific day; in case of non-invasive MV, every day a patient needs non-invasive MV counts as one extra day of MV, irrespective of duration of non-invasive MV that specific day.
Length of Stay in ICU on Day 90 | Until day 90
  Time between admission and discharge or death
Length of Stay in Hospital on Day 90 | Until day 90
  Time between admission and discharge or death
All-cause ICU Mortality | Until day 90
  Any death during ICU stay
All-cause Hospital Mortality | Until day 90
  Any death during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, MD, PhD, Study Chair — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Ary Serpa Neto, MD, MSc, Study Director — PRoVENT Study Trial Coordinator, Department of Intensive Care, Academic Medical Center, University of Amsterdam; Paolo Pelosi, MD, PhD, Principal Investigator — Department of Surgical Sciences and Integrated Diagnostics, University of Genoa, Italy; Marcelo Gama de Abreu, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, University Hospital Carl Gustav Carus, Technical University Dresden, Germany; Carmen SV Barbas, MD, PhD, Principal Investigator — Department of Intensive Care, Hospital Israelita Albert Einstein
Locations (13):
- Medical University Viena, Vienna, Austria
- University Hospital Leuven, Leuven, Belgium
- Brazil (2):
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
- Hospital Clínico de la Pontificia Universidad Católica de Chile, Santiago, Chile
- Saint Eloi University Hospital, Montpellier, France
- Germany (3):
  - University Hospital Bonn, Bonn
  - University Clinic Carl Gustav Carus, Dresden
  - University of Leipzig, Leipzig
- Italy (2):
  - University of Genoa, Genoa
  - University of Insubria, Varese
- Academic Medical Centre, Amsterdam, Netherlands
- Hospital Universitari Germans Trias I Pujol, Barcelona, Spain

REFERENCES:
- [Background] Hemmes SN, Serpa Neto A, Schultz MJ. Intraoperative ventilatory strategies to prevent postoperative pulmonary complications: a meta-analysis. Curr Opin Anaesthesiol. 2013 Apr;26(2):126-33. doi: 10.1097/ACO.0b013e32835e1242. PMID 23385321
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Determann RM, Royakkers A, Wolthuis EK, Vlaar AP, Choi G, Paulus F, Hofstra JJ, de Graaff MJ, Korevaar JC, Schultz MJ. Ventilation with lower tidal volumes as compared with conventional tidal volumes for patients without acute lung injury: a preventive randomized controlled trial. Crit Care. 2010;14(1):R1. doi: 10.1186/cc8230. Epub 2010 Jan 7. PMID 20055989
- [Background] Severgnini P, Selmo G, Lanza C, Chiesa A, Frigerio A, Bacuzzi A, Dionigi G, Novario R, Gregoretti C, de Abreu MG, Schultz MJ, Jaber S, Futier E, Chiaranda M, Pelosi P. Protective mechanical ventilation during general anesthesia for open abdominal surgery improves postoperative pulmonary function. Anesthesiology. 2013 Jun;118(6):1307-21. doi: 10.1097/ALN.0b013e31829102de. PMID 23542800
- [Background] Serpa Neto A, Barbas CSV, Artigas A, et al. Rationale and Study Design of Provent-An International Multicenter Observational Study on Practice of Ventilation in Critically Ill Patients without ARDS. J Clin Trials 2013;3;[in press]
- [Derived] Serafini SC, Cinotti R, Asehnoune K, Battaglini D, Robba C, Neto AS, Pisani L, Mazzinari G, Tschernko EM, Schultz MJ; PRoVENT, the PRoVENT-iMiC and ENIO, investigators. Potentially modifiable ventilation factors associated with outcome in neurocritical care vs. non-neurocritical care patients: Rational and protocol for a patient-level analysis of PRoVENT, PRoVENT-iMiC and ENIO (PRIME). Rev Esp Anestesiol Reanim (Engl Ed). 2025 May;72(5):501690. doi: 10.1016/j.redare.2025.501690. Epub 2025 Feb 15. PMID 39961531
- [Derived] Serafini SC, van Meenen DMP, Pisani L, Neto AS, Ball L, de Abreu MG, Algera AG, Azevedo L, Bellani G, Dondorp AM, Fan E, Laffey JG, Pham T, Tschernko EM, Schultz MJ, van der Woude MCE; ERICC; LUNG SAFE; PRoVENT; PRoVENT-iMiC-investigators. Different ventilation intensities among various categories of patients ventilated for reasons other than ARDS--A pooled analysis of 4 observational studies. J Crit Care. 2024 Jun;81:154531. doi: 10.1016/j.jcrc.2024.154531. Epub 2024 Feb 10. PMID 38341938
- [Derived] Simonis FD, Barbas CSV, Artigas-Raventos A, Canet J, Determann RM, Anstey J, Hedenstierna G, Hemmes SNT, Hermans G, Hiesmayr M, Hollmann MW, Jaber S, Martin-Loeches I, Mills GH, Pearse RM, Putensen C, Schmid W, Severgnini P, Smith R, Treschan TA, Tschernko EM, Vidal Melo MF, Wrigge H, de Abreu MG, Pelosi P, Schultz MJ, Neto AS; PRoVENT investigators; PROVE Network investigators. Potentially modifiable respiratory variables contributing to outcome in ICU patients without ARDS: a secondary analysis of PRoVENT. Ann Intensive Care. 2018 Mar 21;8(1):39. doi: 10.1186/s13613-018-0385-7. PMID 29564726
- [Derived] Neto AS, Barbas CSV, Simonis FD, Artigas-Raventos A, Canet J, Determann RM, Anstey J, Hedenstierna G, Hemmes SNT, Hermans G, Hiesmayr M, Hollmann MW, Jaber S, Martin-Loeches I, Mills GH, Pearse RM, Putensen C, Schmid W, Severgnini P, Smith R, Treschan TA, Tschernko EM, Melo MFV, Wrigge H, de Abreu MG, Pelosi P, Schultz MJ; PRoVENT; PROVE Network investigators. Epidemiological characteristics, practice of ventilation, and clinical outcome in patients at risk of acute respiratory distress syndrome in intensive care units from 16 countries (PRoVENT): an international, multicentre, prospective study. Lancet Respir Med. 2016 Nov;4(11):882-893. doi: 10.1016/S2213-2600(16)30305-8. Epub 2016 Oct 4. PMID 27717861
- See also: PRoVENT website — http://sites.google.com/site/proventtrial/home